CLINICAL TRIAL: NCT00116350
Title: Misoprostol for the Treatment of Primary Postpartum Hemorrhage
Brief Title: Misoprostol for the Treatment of Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Family Care International (Other)
Responsible Party: Gynuity Health Projects, Gynuity Health Projects
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2.4.1; WIRB #20041878/1063615
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; Misoprostol; Developing countries; Maternal morbidity; Randomized controlled trial
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): 800 mcg sublingual misoprostol
  Interventions: Drug: Misoprostol
- Oxytocin (Active Comparator): 40 IU Oxytocin IV
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — 800 mcg sublingual misoprostol
  Arms: Misoprostol
Drug: Oxytocin — 40 IU Oxytocin IV
  Arms: Oxytocin

SUMMARY:
The purpose of this study is to test whether misoprostol is as effective as oxytocin for treating primary postpartum hemorrhage (PPH) with uterine atony as the suspected cause in two circumstances: 1) where women have received prophylactic uterotonics in the third stage of labor; and 2) where no prophylactic uterotonics have been given in the third stage of labor.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) remains a major cause of maternal deaths worldwide. Misoprostol offers several advantages over oxytocin and ergometrine, the drugs currently used to treat PPH. For example, misoprostol is stable at high temperatures and has a shelf life of several years, it is easy to administer, it can be given to hypertensive patients, and it is inexpensive. This randomized, double-blind placebo-controlled trial will test whether misoprostol is as effective as oxytocin in treating primary PPH in hospital births, both when women have received prophylactic uterotonics in the third stage of labor and when they have not.

Blood loss will be measured for all consenting women who deliver vaginally. If PPH occurs and uterine atony is the suspected cause, women will be randomized to receive either: a) four 200 µg pills of misoprostol sublingually and an IV of saline (resembling oxytocin) or b) four placebo tablets resembling misoprostol sublingually and 40 IU oxytocin by IV. This study seeks to answer the following questions:

* Is misoprostol as effective as oxytocin for treatment of primary PPH for women who do and do not receive oxytocin prophylaxis in the third stage of labor?
* Does misoprostol have an acceptable safety profile when given as an 800 µg sublingual dose to treat PPH?
* Is the side effect profile of misoprostol acceptable to women?

This study will take place in hospitals located in Burkina Faso, Ecuador, Egypt, Turkey, and Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery
* Postpartum hemorrhage due to suspected uterine atony
* Depending on study group: administration of prophylactic uterotonics in third stage of labor

Exclusion Criteria:

* Known allergy to misoprostol or other prostaglandin
* C-section for current delivery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1786 (Actual)
Dates: Start 2005-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Need for additional treatment after initial PPH study treatment | all additional interventions recorded following initial uterotonic treatment

SECONDARY OUTCOMES:
Mean blood loss after PPH treatment | blood loss measured for minimum of 1 hour or until active bleeding ceases
Change in hemoglobin from pre-delivery to postpartum | Pe-delivery hemoblogin measured upon entry into labor ward; postpartum Hb measured 12-24 hrs after removal of IV
Time to bleeding cessation | Time to bleeding cessation recorded
Blood transfusion | any blood transfusion recorded after delivery and prior to discharge
Side effects | any observed or reported side effects recorded following treatment and prior to discharge
Acceptability for women | Exit interview conducted prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Jennifer Blum, MPH, Study Director — Gynuity Health Projects; Rasha Dabash, MPH, Study Director — Gynuity Health Projects; Sheila Raghavan, M.Sc., Study Director — Gynuity Health Projects; Ayisha Diop, MPH, Study Director — Gynuity Health Projects; Ilana Dzuba, M.H.Sc., Study Director — Gynuity Health Projects; Jill Durocher, Study Director — Gynuity Health Projects
Locations (6):
- Centre Hospitalier Universitaire Souro Sanou de Bobo Dioulasso, Bobo Diolasso, Burkina Faso
- Hospital Gineco-Obstetrico Isidro Ayora, Quito, Ecuador
- Egypt (2):
  - Alexandria University Hospital, Shatby Maternity Hospital, Alexandria
  - El-Galaa Teaching Hospital, Cairo
- Ministry of Health Ankara Etlik Maternity and Teaching-Research Hospital, Ankara, Turkey (Türkiye)
- Cu Chi Hospital, Tu Du Hospital, Hocmon Hospital, Binh Duong Hospital, Ho Chi Minh City and Binh Duong Province, Vietnam

REFERENCES:
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518
- [Derived] Blum J, Winikoff B, Raghavan S, Dabash R, Ramadan MC, Dilbaz B, Dao B, Durocher J, Yalvac S, Diop A, Dzuba IG, Ngoc NT. Treatment of post-partum haemorrhage with sublingual misoprostol versus oxytocin in women receiving prophylactic oxytocin: a double-blind, randomised, non-inferiority trial. Lancet. 2010 Jan 16;375(9710):217-23. doi: 10.1016/S0140-6736(09)61923-1. Epub 2010 Jan 6. PMID 20060162
- [Derived] Winikoff B, Dabash R, Durocher J, Darwish E, Nguyen TN, Leon W, Raghavan S, Medhat I, Huynh TK, Barrera G, Blum J. Treatment of post-partum haemorrhage with sublingual misoprostol versus oxytocin in women not exposed to oxytocin during labour: a double-blind, randomised, non-inferiority trial. Lancet. 2010 Jan 16;375(9710):210-6. doi: 10.1016/S0140-6736(09)61924-3. Epub 2010 Jan 6. PMID 20060161
- See also: Gynuity Health Projects website — http://www.gynuity.org